CLINICAL TRIAL: NCT02887456
Title: Endodontic Treatment of Primary Teeth Using Mineral Trioxide Aggregate Paste - Protocol of a Phase 2 Randomized Clinical Trial
Brief Title: Endodontic Treatment of Primary Teeth Using Mineral Trioxide Aggregate Paste
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fausto Medeiros Mendes, Associated Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EndoMTA
Record Dates: First submitted 2016-06-14; First posted 2016-09-02 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Teeth, Endodontically-Treated
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitapex (Active Comparator): Endodontic treatment using Vitapex
  Interventions: Drug: Endodontic treatment using Vitapex
- MTA paste (Experimental): Endodontic treatment using MTA paste
  Interventions: Drug: Endodontic treatment using MTA paste

INTERVENTIONS:
Drug: Endodontic treatment using Vitapex — Endodontic treatment using Vitapex
  Arms: Vitapex
Drug: Endodontic treatment using MTA paste — Endodontic treatment using MTA paste
  Arms: MTA paste

SUMMARY:
The maintenance of primary teeth until their exfoliation has been one of the main purposes of Pediatric Dentistry, are they representing the fundamental basis for proper occlusion of the permanent dentition. Often, injuries or extensive dental caries reach the pulp of deciduous teeth making maintenance on these dependent endodontic treatment arc. Thus, this study was to conduct a randomized clinical trial is to evaluate the performance of endodontic treatment in primary teeth using MTA paste, comparing to Vitapex.

DETAILED DESCRIPTION:
After approval by the ethics committee of the patients Faculty of Dentistry, University of São Paulo that having root canal filling of primary teeth will be invited to participate in the study. A clinical examination and prior radiographic diagnosis will be-held. The patient will be randomized to one of two groups and will be made the endodontics by a dentist. The patient will be accompanied with periods of one week, one month and three months by a blinded evaluator. The outcome will be the success or failure of endodontic treatments evaluated through permanent tooth in the arch on clinical and radiographic conditions of normality. The longevity of the treatments will be evaluated by estimating survival rates by Kaplan-Meier. The differences between the survival rates according to the type of proposed endodontic treatment will be analyzed using the log-rank test with a minimum significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Primary teeth with pulp diagnosis and need endodontic treatment
* Patients whose guardians consent to their participation in the survey
* fistula or abscess
* bone rarefaction or visual diagnosis
* teeth in the remaining tooth structure and location of the injury rehabilitation permit do not have internal or external resorption involving more than one third of the root length
* have no bone loss in lateral root and disruption crypt and the presence of at least half of root

Exclusion Criteria:

* health problems systemic
* congenital facial deformities
* facial tumors
* syndromes

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2016-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Success or failure of endodontic treatments | 3 months
  The success or failure of endodontic treatments evaluated by the time spent in the tooth arch in clinical conditions of normality, able to maintain or restore the health of periodical tissues after the treatment. Clinical criteria for determining success are: absence of fistula, absence of painful symptoms and pathological absence of adequate mobility and gingival contour. Radiographically, the success criteria are: absence / reduction of periapical bone rarefaction in anterior and absence / bone rarefaction in the furcation area of later, maintaining the periradicular space, root resorption compatible with the eruptive phase and absence of pathological bone resorption. To evaluate the reduction of lesions or appearance of new lesions will be between the initial and follow-up radiographs. Radiographs will be scanned and the end of the bone rarefactions starting area and will be measured on a software image analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Carmela Bresolin, Principal Investigator — Faculdade de Odontologia da USP
Locations (1):
- Carmela Bresolin, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garcia-Godoy F. Evaluation of an iodoform paste in root canal therapy for infected primary teeth. ASDC J Dent Child. 1987 Jan-Feb;54(1):30-4. PMID 3468139
- [Background] Rifkin A. A simple, effective, safe technique for the root canal treatment of abscessed primary teeth. ASDC J Dent Child. 1980 Nov-Dec;47(6):435-41. No abstract available. PMID 6934178
- [Background] Mello-Moura AC, Fanaro J, Nicoletti MA, Mendes FM, Wanderley MT, Guedes-Pinto AC. Variability in the proportion of components of iodoform-based Guedes-Pinto paste mixed by dental students and pediatric dentists. Indian J Dent Res. 2011 Nov-Dec;22(6):781-5. doi: 10.4103/0970-9290.94668. PMID 22484870
- [Background] Cerqueira DF, Mello-Moura AC, Santos EM, Guedes-Pinto AC. Cytotoxicity, histopathological, microbiological and clinical aspects of an endodontic iodoform-based paste used in pediatric dentistry: a review. J Clin Pediatr Dent. 2008 Winter;32(2):105-10. doi: 10.17796/jcpd.32.2.k1wx5571h2w85430. PMID 18389674
- [Background] Amorim Lde F, Toledo OA, Estrela CR, Decurcio Dde A, Estrela C. Antimicrobial analysis of different root canal filling pastes used in pediatric dentistry by two experimental methods. Braz Dent J. 2006;17(4):317-22. doi: 10.1590/s0103-64402006000400010. PMID 17262146
- [Background] Mass E, Zilberman UL. Endodontic treatment of infected primary teeth, using Maisto's paste. ASDC J Dent Child. 1989 Mar-Apr;56(2):117-20. PMID 2656788
- [Result] Nurko C, Ranly DM, Garcia-Godoy F, Lakshmyya KN. Resorption of a calcium hydroxide/iodoform paste (Vitapex) in root canal therapy for primary teeth: a case report. Pediatr Dent. 2000 Nov-Dec;22(6):517-20. PMID 11132515
- [Result] Kopel HM. Root canal therapy for primary teeth. J Mich State Dent Assoc. 1970 Feb;52(2):28-33 passim. No abstract available. PMID 5263926
- [Result] George S, Anandaraj S, Issac JS, John SA, Harris A. Rotary endodontics in primary teeth - A review. Saudi Dent J. 2016 Jan;28(1):12-7. doi: 10.1016/j.sdentj.2015.08.004. Epub 2015 Nov 22. PMID 26792964
- [Result] Wong AW, Tsang CS, Zhang S, Li KY, Zhang C, Chu CH. Treatment outcomes of single-visit versus multiple-visit non-surgical endodontic therapy: a randomised clinical trial. BMC Oral Health. 2015 Dec 19;15:162. doi: 10.1186/s12903-015-0148-x. PMID 26687126
- [Result] Moskovitz M, Tickotsky N, Ashkar H, Holan G. Degree of root resorption after root canal treatment with iodoform-containing filling material in primary molars. Quintessence Int. 2012 May;43(5):361-8. PMID 22536587
- [Result] Mortazavi M, Mesbahi M. Comparison of zinc oxide and eugenol, and Vitapex for root canal treatment of necrotic primary teeth. Int J Paediatr Dent. 2004 Nov;14(6):417-24. doi: 10.1111/j.1365-263X.2004.00544.x. PMID 15525310